CLINICAL TRIAL: NCT03730376
Title: Patient and Consumer Decision Making in a Hypothetical Case of Carpal Tunnel Syndrome
Brief Title: Decision Making in Hypothetical Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Robin Kamal, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 47392, 47580
Record Dates: First submitted 2018-11-02; First posted 2018-11-05 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into 1 of 2 study arms arm 1: control arm 2: intervention.
  We will use a random block generator to assign participants to their study arm.
Who Masked: Participant, Care Provider
Masking Description: The care provider and patient will not be informed as to which group the participant is in
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants in the control group will be given a hypothetical scenario about carpal tunnel syndrome and asked to make a treatment decision for that hypothetical patient.
- Intervention (Experimental): Participants in the intervetion group will be given a hypothetical scenario about carpal tunnel syndrome as well as information about the cost of treatment and asked to make a treatment decision for that hypothetical patient.
  Interventions: Other: Cost Information

INTERVENTIONS:
Other: Cost Information — participants will be given information on the personal and societal costs
  Arms: Intervention

SUMMARY:
Participants will be presented with a hypothetical scenario of carpal tunnel and asked to make a decision for that case.

DETAILED DESCRIPTION:
Participants will be randomized into 1 of 2 groups and receive a hypothetical scenario of carpal tunnel, with or without cost information, and asked to decide if that hypothetical patient should undergo a carpal tunnel release.

ELIGIBILITY:
Inclusion Criteria:

* patients presenting to hand clinic OR mturk workers
* age 18 or older

Exclusion Criteria:

* traumatic mechanism of injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Decision to have Treatment | immediately after completing survey
  Participants are asked to answer "Should you get surgery right now," with the options of definitely yes, probably, maybe, maybe not, probably not, and definitely not

SECONDARY OUTCOMES:
Opinion on healthcare costs | immediately after completing survey
  a 7 item, likert response questionnaire used to elicit participant opinions on cost in health care. This is a non-validated tool.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Health Care, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No